CLINICAL TRIAL: NCT00845858
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Dose-Ranging Clinical Study to Evaluate the Efficacy and Safety of Metoclopramide Nasal Spray Solution in Diabetic Subjects With Gastroparesis
Brief Title: Efficacy and Safety of Metoclopramide Nasal Spray Solution in Diabetic Patients With Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evoke Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METO-IN-002
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-11

CONDITIONS: Gastroparesis; Diabetic Gastroparesis; Diabetes; Diabetes Mellitus; Delayed Gastric Emptying
Keywords: Gastroparesis; Diabetic Gastroparesis; Diabetes; Diabetes Mellitus; Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metoclopramide Nasal Spray 10 mg (Active Comparator)
  Interventions: Drug: metoclopramide
- Metoclopramide Nasal Spray 14 mg (Active Comparator)
  Interventions: Drug: metoclopramide
- Placebo Nasal Spray (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metoclopramide — 30 minutes before meals and at bedtime for 4 weeks
  Other Names: Reglan
  Arms: Metoclopramide Nasal Spray 10 mg; Metoclopramide Nasal Spray 14 mg
Drug: Placebo — 30 minutes before meals and at bedtime
  Arms: Placebo Nasal Spray

SUMMARY:
To evaluate the safety and the effectiveness of two doses of metoclopramide nasal spray solution, 10 mg and 14 mg, compared to placebo in reducing the symptoms of diabetic gastroparesis.

ELIGIBILITY:
Inclusion Criteria

1. Male subjects and non-pregnant, non-lactating female subjects between the ages of 18 and 75 years (inclusive)
2. Willing and able to give written informed consent to participate in the study
3. Ability to read and understand English
4. Diagnosis of Type 1 or Type 2 diabetes
5. Diagnosis of diabetic gastroparesis previously documented
6. A mean daily GCSI-DD score of ≥2 and ≤4 for the 7 days prior to the Randomization Visit (Visit 3, Day 0)
7. Female subjects of childbearing potential, defined as not surgically sterile or at least 2 years postmenopausal, must agree to use one of the following forms of contraception from Screening through the last dose of study drug: hormonal (oral, implant, or injection) begun >30 days prior to screening, barrier (condom, diaphragm, or cervical cap with spermicide), intrauterine device (IUD), or vasectomized partner (6-months minimum)
8. No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results (with the exception of lipid profile, glucose and hemoglobin A1c) during screening which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results
9. Willingness to discontinue current treatment for diabetic gastroparesis and to avoid all medications specified by the protocol for the duration of the study

Exclusion Criteria

1. Gastric bypass and gastric banding, gastric pacemakers, post-surgical causes of gastroparesis and disorders known to be associated with abnormal gastrointestinal motility such as active gastric ulcer, active duodenal ulcer, active severe gastritis, gastric cancer, amyloidosis, neuromuscular diseases (including Parkinson's disease), collagen vascular diseases, alcoholism, uremia, malnutrition, and untreated hypothyroidism
2. A history of allergic or adverse responses, including, but not limited to, acute dystonic reactions and tardive dyskinesia to metoclopramide or any comparable or similar product
3. History of or physical findings suggestive of tardive dyskinesia
4. Currently using and unwilling or unable to stop any medication known to be associated with tardive dyskinesia (See Study Reference Manual) prior to Washout (Visit 2)
5. History of allergy to any of the ingredients in the study drug formulation; metoclopramide, citric acid, sodium citrate, benzalkonium chloride, EDTA, or sorbitol
6. History of organ transplant, chronic pancreatitis, gross malabsorptive syndromes, celiac disease, or inflammatory bowel disease
7. Malignancy (with the exception of basal cell carcinoma of the skin) currently present, initially diagnosed or recurring within 5 years of enrollment
8. History of other clinically significant renal, hepatic, neurologic, hematologic, oncologic, pulmonary, psychiatric, cardiovascular or infectious disease, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results
9. Have renal dysfunction calculated as creatinine clearance (CrCl) < 40 mL/min at Screening (Visit 1)
10. Have a hemoglobin A1c > 12.5% at Screening (Visit 1)
11. Inability or unwillingness to stop using the following agents for 7 days during the Washout Period (Day -7 to Day -1) prior to Randomization (Visit 3, Day 0) and refrain from their use for the 4-week study period; oral and parenteral formulations of metoclopramide, domperidone, tricyclic antidepressants, macrolide antibiotics, prokinetic agents, cholinergic agents, agents with significant anticholinergic effects, narcotic analgesics, orally administered β agonists, spasmolytics, dopamine agonists, monoamine oxidase inhibitors, herbal supplements, fiber or bulking products, and laxatives
12. Use of neurotoxins (e.g., botulinum type A or B) as a treatment for gastroparesis or delayed gastric emptying within 6 months of Screening (Visit 1)
13. Clinically significant abnormal finding or a QTc interval >450 milliseconds (msec) on ECGs obtained at Screening (Visit 1) OR pre- or post-dose at Randomization (Visit 3)
14. Inability or unwillingness to stop using medications associated with Torsades de Pointes or a prolonged QT interval for 30 days prior to the initial symptom assessment and refrain from their use for the 4-week study period (see Study Reference Manual)
15. Female subjects who are trying to conceive, are pregnant, or are lactating
16. Positive serum human chorionic gonadotropin (HCG) pregnancy test at Screening or a positive HCG urine test on Day 0 prior to administration of study drug for women of childbearing potential
17. History of alcohol or drug abuse within the year prior to the Screening Visit, or current known evidence of substance dependence or abuse
18. Participation in a clinical (investigational) trial or receipt of a non-FDA approved therapy within 30 days prior to the Screening Visit (Visit 1) with the exception of domperidone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (65):
  - Digestive Specialists of the Southeast, Dothan, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Desert Sun Gastroenterology, Tucson, Arizona
  - Clopton Clinic, Jonesboro, Arkansas
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Robert M. Karns, MD, a Medical Corporation, Beverly Hills, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Impact Clinical Trials, Los Angeles, California
  - Prime-Care Clinical Research, Mission Viejo, California
  - Infosphere Clinical Research, Inc., West Hills, California
  - Westlake Medical Research, Westlake Village, California
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - AppleMed Research, Inc., Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Newton Medical Center, Conyers, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Saint John's Research Institute, Anderson, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Professional Research Network of Kansas, Wichita, Kansas
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Maryland Digestive Disease Research, LLC, Laurel, Maryland
  - Endoscopic Microsurgery Associates, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Plymouth Clinic, Plymouth, Minnesota
  - CRC of Jackson, LLC, Jackson, Mississippi
  - Gastrointestional Associates, Jackson, Mississippi
  - Digestive Health Specialists, Tupelo, Mississippi
  - Kansas City Gastroenterology & Hepatology, Kansas City, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Medex Healthcare Research, Inc., New York, New York
  - Research Associates of New York, New York, New York
  - Gastroenterology Associates, Poughkeepsie, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - LeBauer Research Associates, Greensboro, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hanover Medical Specialists, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - AGA, Akron, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - PMA Medical Specialists, Limerick, Pennsylvania
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - Medical Specialty Clinic Research, Jackson, Tennessee
  - Holston Medical Group, PC, Kingsport, Tennessee
  - Lovelace Scientific Resources, Austin, Texas
  - Jacinto Medical Group, Baytown (Houston), Texas
  - Dynamed Clinical Research, Houston, Texas
  - Digestive Health Associates of Texas, P.A., Plano, Texas
  - Theda Oaks Endoscopy Center, San Antonio, Texas
  - Trinity Health Care, Tyler, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Gastroenterology, Ltd., Virginia Beach, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Parkman HP, Carlson MR, Gonyer D. Metoclopramide Nasal Spray Reduces Symptoms of Gastroparesis in Women, but not Men, With Diabetes: Results of a Phase 2B Randomized Study. Clin Gastroenterol Hepatol. 2015 Jul;13(7):1256-1263.e1. doi: 10.1016/j.cgh.2014.12.030. Epub 2015 Jan 7. PMID 25576687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoclopramide Nasal Spray 10 mg | Metoclopramide Nasal Spray 14 mg | Placebo Nasal Spray
Started | 96 (95 subjects received allocated intervention. 1 subject withdrew consent and was not dosed.) | 96 (95 subjects received allocated intervention. 1 subject was not eligible and was not dosed.) | 95
Completed | 88 | 84 | 87
Not Completed | 8 | 12 | 8
Not completed — Withdrawal by Subject | 5 | 1 | 1
Not completed — Adverse Event | 3 | 8 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — not eligible | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Provides at least 80% power (alpha=0.05 two sided) to detect a mean difference between treatment groups of 0.5, for the GCSI-DD total score. Based on the literature, the standard deviation (SD) of the endpoint is approximately 1.1 resulting in a sample size of 77 per treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide Nasal Spray 10 mg | Metoclopramide Nasal Spray 14 mg | Placebo Nasal Spray | Total
Number analyzed (Participants) | 96 | 96 | 95 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (12.13) | 50.3 (12.40) | 52.4 (10.03) | 51.4 (11.56)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 81 | 83 | 85 | 249
  >=65 years | 15 | 13 | 10 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 70 | 68 | 203
  Male | 31 | 26 | 27 | 84
Region of Enrollment [Number; unit: participants]
  United States | 96 | 96 | 95 | 287

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is the Change From Baseline to Week 4 of the Treatment Period in the Modified Gastroparesis Cardinal Symptom Index-Daily Diary (mGCSI-DD) Total Score.
Description: Change from Baseline to Week 4 of the treatment period in the mGCSI-DD total score in male and female subjects receiving metoclopramide nasal spray versus subjects receiving placebo.
  The mGCSI-DD is a patient reported outcome measure of gastroparesis symptom severity composed of 4 individual symptoms (listed below) with each symptom graded on a scale from 0 (none) to 5 (very severe).
  1. Nausea (feeling sick to your stomach as if you were going to vomit or throw up)
  2. Early satiety (not able to finish a normal sized meal)
  3. Bloating (feeling like you need to loosen clothes)
  4. Upper abdominal pain (above the navel) The mGCSI-DD daily score is a mean of the 4 individual symptom scores. The total score is a mean of the daily scores for the observation period.
  A mean change (improvement) of >1 category (for example, moderate to mild or severe to moderate) is considered to be clinically meaningful.
Time Frame: 4 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metoclopramide Nasal Spray 10 mg | Metoclopramide Nasal Spray 14 mg | Placebo Nasal Spray
Number analyzed (Participants) | 96 | 96 | 95
units on a scale | -1.2 (1.18) | -1.2 (0.94) | -1.0 (0.89)

2. Other Pre Specified Outcome: The Pre-specified Endpoint is the Change From Baseline to Week 4 of the Treatment Period in the Modified Gastroparesis Cardinal Symptom Index-Daily Diary (mGCSI-DD) Total Score by Gender.
Description: Change from Baseline to Week 4 of the treatment period in the mGCSI-DD total score in Female subjects receiving metoclopramide nasal spray versus Female subjects receiving placebo.
  The mGCSI-DD is a patient reported outcome measure of gastroparesis symptom severity composed of 4 individual symptoms (listed below) with each symptom graded on a scale from 0 (none) to 5 (very severe).
  1. Nausea (feeling sick to your stomach as if you were going to vomit or throw up)
  2. Early satiety (not able to finish a normal sized meal)
  3. Bloating (feeling like you need to loosen clothes)
  4. Upper abdominal pain (above the navel) The mGCSI-DD daily score is a mean of the 4 individual symptom scores. The total score is a mean of the daily scores for the observation period.
  A mean change (improvement) of >1 category (for example, moderate to mild or severe to moderate) is considered to be clinically meaningful.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Female-Metoclopramide Nasal Spray 10 mg; Female-Metoclopramide Nasal Spray 14 mg: metoclopramide: 30 minutes before meals and at bedtime for 4 weeks
- Female-Placebo Nasal Spray: Placebo: 30 minutes before meals and at bedtime
Arm/Group | Female-Metoclopramide Nasal Spray 10 mg | Female-Metoclopramide Nasal Spray 14 mg | Female-Placebo Nasal Spray
Number analyzed (Participants) | 65 | 70 | 68
units on a scale | -1.2 (1.18) | -1.3 (0.98) | -0.8 (0.79)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) (from signing of Informed Consent Form until termination of study drug [28 days]), whether observed by the Investigator, reported by the subject, from laboratory findings, or other means, were captured.
Description: All AEs were followed in accordance with good medical practice until resolved or fully characterized. AEs that were ongoing at the end of the study were followed for at least 72 hours to determine the status of the event.
  All serious and related AEs that occurred within 30 days after the last dose of study drug were captured.
Arm/Group | Metoclopramide Nasal Spray 10 mg | Metoclopramide Nasal Spray 14 mg | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/95 | 2/95 | 3/95
Other Adverse Events (participants affected / at risk) | 53/95 | 57/95 | 53/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide Nasal Spray 10 mg (N=95) | Metoclopramide Nasal Spray 14 mg (N=95) | Placebo Nasal Spray (N=95)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide Nasal Spray 10 mg (N=95) | Metoclopramide Nasal Spray 14 mg (N=95) | Placebo Nasal Spray (N=95)
Dysguesia (Nervous system disorders) | 12 (13) | 13 (14) | 4 (4)
Headache (Nervous system disorders) | 12 (13) | 13 (14) | 11 (13)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 9 (9)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4)
Dyspesia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 5 (5) | 6 (7) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (General disorders) | 1 (1) | 3 (3) | 1 (1)
Hypoglycemia (General disorders) | 1 (1) | 3 (5) | 1 (1)
Decreased Appetite (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Blood Glucose Increase (Investigations) | 0 (0) | 1 (1) | 2 (2)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Glycosylated Haemoglobin Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Pollakiurua (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less